CLINICAL TRIAL: NCT02177409
Title: A Prospective Randomized Open-Label, Blinded-Endpoint (PROBE) Trial Comparing MICARDIS® (Telmisartan) (80 mg QD) and Amlodipine (5 mg QD) in Patients With Mild-to-Moderate Hypertension Using Ambulatory Blood Pressure Monitoring.
Brief Title: Telmisartan Versus Amlodipine in Patients With Mild-to-Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.258
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

ARMS (2):
- Telmisartan (Experimental): 4-week placebo run-in, 8-week fixed dose period
  Interventions: Drug: Telmisartan; Drug: Placebo
- Amlodipine (Active Comparator): 4-week placebo run-in, 8-week fixed dose period
  Interventions: Device: Amlodipine; Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan
Device: Amlodipine
  Arms: Amlodipine
Drug: Placebo

SUMMARY:
The primary aim of the trial is the effect of telmisartan versus amlodipine in lowering ambulatory diastolic and/or systolic blood pressures in the last six hours of the dosing interval in patients with mild-to-moderate hypertension as measured by ambulatory blood pressure monitoring (ABPM)

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate hypertension defined as a mean seated diastolic blood pressure (BP) of ≥ 95 mm Hg and ≤ 114 mm Hg, measured by manual cuff sphygmomanometer, on the last visit (Visit 6) of the four-week placebo run-in period (baseline BP)
* Mean seated systolic blood pressure ≥ 140 mm Hg and ≤ 200 mm Hg, measured by manual cuff at Visit 6 (baseline BP)
* A 24-hour mean ABPM measurement of ≥ 130/85 mm Hg evaluated at Visit 7 (baseline ABPM)
* Age 18 or older
* Ability to provide written informed consent

Exclusion Criteria:

* Pre-menopausal women (last menstruation ≤ 1 year prior to start of screening):

  * who are not surgically sterile (hysterectomy, tubal ligation)
  * who are NOT practicing acceptable means of birth control or who do NOT plan to continue using an acceptable method throughout the study
* Any women:

  * Who has a positive serum pregnancy test at screening (Visit 1) or baseline (Visit 7)
  * Who is nursing
* Hepatic and/or renal dysfunction as defined by the following laboratory parameters

  * SGPT (ALT) (serum glutamate pyruvate transaminase) or SGOT (AST) (serum glutamate oxaloacetate transaminase) greater than two times the upper limit of normal
  * Serum creatinine > 2.3 mg/dL
* At screening (Visit 1): clinically relevant sodium depletion, hyperkalemia, or hypokalemia
* Known or suspected secondary hypertension
* Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; post-renal transplant patients, presence of only one functioning kidney
* Congestive heart failure (CHF) (NYHA (New York Heart Association) class CHF III-IV)
* Unstable angina within the past three months
* Stroke within the past six months
* Myocardial infarction or cardiac surgery within the past three months
* PTCA (percutaneous transluminal coronary angioplasty) within the past three months
* History of angioedema
* Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator
* Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
* Administration of digoxin or other digitalis-type drugs
* Patients with insulin-dependent diabetes mellitus whose diabetes has not been stable and controlled for at least the past three months as defined by an HbA1C ≥ 10%
* Known drug or alcohol dependency within the past one year period
* Concomitant administration of medications known to affect blood pressure, except medications allowed by the protocol
* Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 AM (ante meridian)
* Patients receiving any investigational therapy within one month of signing the informed consent form. Note that patients who have participated in previous MICARDIS (telmisartan) studies may participate in this study provided there has been at least one month between discontinuing the previous study and signing the consent for the present study
* Known hypersensitivity to any component of the formulations
* Any clinical condition which, in the opinion of the investigator would not allow safe completion of the protocol and safe administration of trial medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 1998-04; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in diastolic and systolic blood pressure during the last six hours of a 24-hour dosing interval, measured by ambulatory blood pressure monitoring | Baseline (day 1), day 57 of the open-label period

SECONDARY OUTCOMES:
Changes from baseline in diastolic and systolic blood pressure during other times during the 24-hour ABPM profile | Baseline (day 1), up to day 57 of the open-label period
Changes from baseline in seated trough diastolic and systolic blood pressures as measured by manual cuff | Baseline (day 27 of the single-blind period), days 1, 14, 28, 56 and 57 of the open-label period
Blood pressure responder rates based on ABPM | day 56 and 57 of the open-label period
Blood pressure responder rates based on manual cuff measurements | days 14, 28, 56 and 57 of the open-label period